CLINICAL TRIAL: NCT04197505
Title: Application of Forward-looking Infrared for the Identification and Evaluation of Fractures in the Acute Trauma Setting
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Lost funding due to COVID-19
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 19-01424
Record Dates: First submitted 2019-12-11; First posted 2019-12-13 (Actual); Last update posted 2021-10-11 (Actual); Status verified 2021-10

CONDITIONS: Acute Fracture

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Acute fracture specific (Experimental): The FLIR E95 camera will be used for the study. The injured extremity will be scanned with the thermal camera and a second scan will be performed on the non-injured extremity to provide an internal control for any differences in room temperature and humidity. Prior to scanning, both the injured and non-injured extremity will remain uncovered for 10 minutes, about the length of an average office visit, and the areas to be scanned will remain free from contact by the patient or interviewer during this time period. The camera will be held 2 feet away from the extremity at a 90º angle to limit reading contamination from objects other than the patient.
  Interventions: Behavioral: FLIR E95 camera

INTERVENTIONS:
Behavioral: FLIR E95 camera — Video will be recorded during the thermal reading for later computer analysis. The following variables will be analyzed: (1) the difference between the mean temperature between the injured and healthy extremities, (2) the difference between the maximum temperatures of both the injured and healthy extremities (ΔTmax), and (3) the difference between the area covered by each isotherm in both the injured and uninjured extremities (Δpix). FLIR software tools and MATLAB software will be used for the analysis.

SUMMARY:
The overall objective of this study is to (1) determine whether thermal imaging can be used during an acute trauma patient's secondary or tertiary survey to identify injury sites with an underlying fracture, and to (2) investigate whether thermal imaging can predict those patients whose fractures will result in a non-union.

DETAILED DESCRIPTION:
Human subjects will be enrolled into the study from NYU Langone Health and Bellevue Hospital Center. When orthopaedic surgery is consulted for management of a fracture, the patient will be offered enrollment into the study. The collected data will be assigned a letter and number associated for references with the patient's age, type of fracture, and time since original injury to thermal imaging scan. If any patient receives a thermal imaging scan at their initial injury evaluation, then he or she will also receive thermal imaging scans at all follow-up appointments to track changes in temperature over the healing process. No obtunded or unresponsive patients will be enrolled into the study. The goal will be to have to thirty patients enrolled into both acute fracture and non-union arms of the proposal for a total of sixty subjects. Age, gender, ethnicity, smoking status, medical history, and surgical history will be recorded for future confounding analysis.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged 18 to 95
* Have fracture injury

Exclusion Criteria:

* Subjects suffering from a hypothermia- or hyperthermia - related illness or other environmental exposure-type illness
* Those with a concomitant fracture
* Subjects with no specific medical history or surgical history
* Subjects who cannot provide informed consent

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-01 (Estimated); Primary Completion 2024-07 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
Comparison of thermal imaging of extremity with and without fracture | through study completion, an average of 18 months
  The FLIR E95 thermal imaging camera will be used to obtain a temperature evaluation of the injury site. The extremity with the underlying fracture will have a higher temperature reading when compared to the contralateral extremity without a fracture. Thermal imaging was selected for the proposed work due to its feasibility and potential to be a useful tool in the acute trauma setting. A thermal imaging camera detects infrared radiation and converts it to visible light. The FLIR E95 utilizes a class two laser with an output power below 1mW and this laser is considered safe without a skin or materials burn hazard unless a person deliberately stares into the beam

SECONDARY OUTCOMES:
Change in thermal imaging predicting non-union | through study completion, an average of 18 months
  Using the FLIR E95 thermal imaging camera, to monitor progression of fracture healing and identify patients proceeding towards a non-union. A fracture proceeding towards a non-union will have a persistently higher local temperature compared to an appropriately healing fracture. Thermal imaging was selected for the proposed work due to its feasibility and potential to be a useful tool in the acute trauma setting. A thermal imaging camera detects infrared radiation and converts it to visible light. The FLIR E95 utilizes a class two laser with an output power below 1mW and this laser is considered safe without a skin or materials burn hazard unless a person deliberately stares into the beam

CONTACTS AND LOCATIONS:
Overall Officials: Philipp Leucht, Principal Investigator — NYU Langone

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data.Upon reasonable request. Requests should be directed to john.dankert@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.